CLINICAL TRIAL: NCT01362296
Title: A Phase II, Open-label, Multicenter, Randomized Study to Assess the Efficacy and Safety of GSK1120212 Compared With Docetaxel in 2nd Line Subjects With Targeted Mutations (KRAS, NRAS, BRAF, MEK1) in Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC Stage IV)
Brief Title: An Open-label Study of GSK1120212 Compared With Docetaxel in Stage IV KRAS-mutant Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114653
Record Dates: First submitted 2011-05-19; First posted 2011-05-30 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-06

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: NRAS; docetaxel; NSCLC; GSK1120212; MEK inhibitor; targeted therapy; KRAS; BRAF
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — trametinib; Docetaxel

ARMS (2):
- GSK1120212 (Experimental): Oral once daily
  Interventions: Drug: GSK1120212
- docetaxel (Active Comparator): IV once every 3 weeks
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: GSK1120212 — Oral once daily
  Arms: GSK1120212
Drug: docetaxel — IV once every 3 weeks
  Arms: docetaxel

SUMMARY:
This is a phase II, open-label, multicenter, randomized study to evaluate the efficacy and safety of GSK1120212 compared with docetaxel in the second line setting for subjects with locally advanced or metastatic (Stage IV) Non-small cell lung cancer (NSCLC) harboring a KRAS mutation who have failed one platinum-containing chemotherapy regimen. A small subset of NSCLC subjects harboring BRAF, NRAS, or MEK1 mutations will be randomized in addition to the primary KRAS population, for exploratory purposes.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old with histologically- or cytologically-confirmed diagnosis of adenocarcinoma Stage IV NSCLC with a positive mutational status for the KRAS, NRAS, BRAF, or MEK1 gene.
* Documented tumor progression after receiving at least one, but not more than one, prior approved platinum-containing chemotherapy regimen for advanced stage/metastatic NSCLC.
* Measurable disease per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Performance status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Life expectancy of at least three months in the opinion of the investigator.
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of randomization to study treatment and agree to use effective contraception. Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from the time of randomization to study medication until at least four weeks after the last dose of study treatment.
* Adequate baseline organ function.

Exclusion Criteria:

* History of another malignancy.
* Any serious and/or unstable pre-existing medical disorder, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Treatment with a BRAF or MEK inhibitor or docetaxel as monotherapy or as part of a combination regimen.
* Anti-cancer therapy (including chemotherapy and radiation therapy) within the last three weeks.
* History or current evidence / risk of retinal vein occlusion or central serous retinopathy.
* Any current or history of tumor manifestation in the Central Nervous System.
* History or evidence of cardiovascular risk, including QTcB >=480 msec, uncontrolled arrhythmias, acute coronary syndrome, coronary angioplasty, or stenting within 6 months prior to randomization, >=Class II congestive heart failure, treatment refractory hypertension, intra-cardiac defibrillators or permanent pacemakers or cardiac metastases.
* Known Human Immunodeficiency Virus, Hepatitis B Virus (HBV), or Hepatitis C Virus (HBC) infection (with the exception of chronic or cleared HBV and HCV infection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (48):
- United States (23):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Athens, Georgia
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Vancouver, Washington
- France (5):
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Villejuif
- Greece (4):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Neo Faliro
  - GSK Investigational Site, Thessaloniki
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Törökbálint
- Italy (2):
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
- Netherlands (5):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Zwolle
- GSK Investigational Site, Seoul, South Korea
- Spain (5):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Pamplona

REFERENCES:
- [Derived] Blumenschein GR Jr, Smit EF, Planchard D, Kim DW, Cadranel J, De Pas T, Dunphy F, Udud K, Ahn MJ, Hanna NH, Kim JH, Mazieres J, Kim SW, Baas P, Rappold E, Redhu S, Puski A, Wu FS, Janne PA. A randomized phase II study of the MEK1/MEK2 inhibitor trametinib (GSK1120212) compared with docetaxel in KRAS-mutant advanced non-small-cell lung cancer (NSCLC)dagger. Ann Oncol. 2015 May;26(5):894-901. doi: 10.1093/annonc/mdv072. Epub 2015 Feb 26. PMID 25722381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met eligibility criteria at Screening were then randomized to the treatment period. A total of 134 participants were randomized, and 130 participants entered the treatment period.
Pre-assignment Details: In the Randomized Phase (RP), participants were treated until disease progression (PD), death, or unacceptable adverse events were experienced. After PD in the RP, participants were given the option of crossing over to the alternative treatment arm in a Cross-over Phase (CP).
Groups:
- GSK1120212 2 mg in RP; GSK1120212 2 mg in CP: Participants received GSK1120212 2 milligrams (mg) orally once daily continuously in the Randomized Phase (RP). Participants continued treatment until disease progression, death, or unacceptable adverse events were experienced. Participants who experienced disease progression in the RP were given the option of crossing over to the alternative treatment arm (docetaxel 75 milligrams per meters squared [mg/m^2]), and continuing in the Cross-over Phase (CP).
- Docetaxel 75 mg/m^2 in RP; Docetaxel 75 mg/m^2 in CP: Participants received docetaxel 75 mg per meters squared (m^2) intravenously (IV) every 3 weeks in the RP. Participants continued treatment on a 21-day cycle until disease progression, death, or unacceptable adverse events were experienced. Participants who experienced disease progression in the RP were given the option of crossing over to the alternative treatment arm (GSK1120212 2 mg), and continuing in the CP.
Period: Randomized Phase (RP)
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP | GSK1120212 2 mg in CP | Docetaxel 75 mg/m^2 in CP
Started | 87 | 43 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 87 | 43 | 0 | 0
Not completed — PD including Death due to PD | 56 | 28 | 0 | 0
Not completed — Physician Decision | 1 | 9 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Adverse Event | 20 | 4 | 0 | 0
Not completed — Study Closed/Terminated | 8 | 1 | 0 | 0
Period: Crossover Phase
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP | GSK1120212 2 mg in CP | Docetaxel 75 mg/m^2 in CP
Started | 0 (These participants elected to enter the Crossover Phase at the time of disease progression.) | 0 (These participants elected to enter the Crossover Phase at the time of disease progression.) | 23 (These participants elected to enter the Crossover Phase at the time of disease progression.) | 2 (These participants elected to enter the Crossover Phase at the time of disease progression.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 23 | 2
Not completed — PD including Death due to PD | 0 | 0 | 16 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 4 | 0
Not completed — Study Closed/Terminated | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP | Total
Number analyzed (Participants) | 89 | 45 | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (8.97) | 60.9 (10.06) | 61.2 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 22 | 65
  Male | 46 | 23 | 69
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 73 | 32 | 105
  Asian - East Asian Heritage | 11 | 9 | 20
  White - Arabic/North African Heritage | 1 | 3 | 4
  African American/African Heritage | 3 | 0 | 3
  Asian - South East Asian Heritage | 0 | 1 | 1
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Assessed by the Investigator (INV)
Description: PFS is defined as the time from RAN until the earliest date of documented radiological PD or DT due to any cause. PD was assessed by the INV according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. PD is defined as at least a 20% increase in the sum of the diameters (SD) of target lesions with an absolute increase of at least 5 millimeters (mm) or the appearance of at least 1 new lesion, or the worsening of non-target lesions significant enough to require study treatment discontinuation. For participants (PAR) who did not have a documented date of PD or DT, PFS was censored at the date of the last adequate assessment. For PAR who received subsequent anti-cancer therapy prior to the date of documented PD or DT, PFS was censored at the date of the last adequate assessment prior to the initiation of therapy.
Time Frame: From randomization (RAN) until the earliest date of documented radiological disease progression (PD) or death (DT) due to any cause (maximum of 10.2 months)
Population: Modified Intent-to-Treat (MITT) Population: all randomized participants with KRAS mutation-positive non-small cell lung cancer (NSCLC), whether or not treatment was administered
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP
Number analyzed (Participants) | 86 | 43
Weeks | 11.7 [7.0 to 12.4] | 11.4 [6.1 to 18.3]
Statistical Analysis 1: Comparison: GSK1120212 2 mg in RP vs Docetaxel 75 mg/m^2 in RP; Test type: Superiority or Other; p = 0.5197, Log Rank — P-value from the stratified log-rank was adjusted for gender (male versus female); Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.75 to 1.75] — HRs were estimated using a Pike estimator. The HR from the stratified log-rank test was adjusted for gender (male versus female)

2. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline in the Indicated Clinical Chemistry Parameters: Randomized Phase
Description: Clinical chemistry parameters were summarized according to National Cancer Institutes (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade, version 4.0. Grade (G) 1, Mild; Grade 2, Moderate; Grade 3 (G3), Severe; Grade 4 (G4), Life-threatening or disabling; Grade 5, Death. Data are presented for only those parameters for which an increase to any G, G3, or G4 occurred. Clinical chemistry parameters included: albumin, alkaline phosphatase (ALKP), alanine amino transferase (ALT), aspartate amino transferase (AST), total bilirubin, calcium (hypercalcemia), calcium (hypocalcemia), creatine kinase, creatinine, glucose (hyperglycemia), glucose (hypoglycemia), potassium (hyperkalemia), potassium (hypokalemia), sodium (hypernatremia), and sodium (hyponatremia). Worst-case on-therapy changes from Baseline were summarized. Worst-case on-therapy was defined using the on-therapy window and changes were indentified using both scheduled and unscheduled assessments.
Time Frame: Baseline; Days 1, 8, and 15 of Cycle 1; and Day 1 of every cycle thereafter until treatment discontinuation of the Randomized Phase (up to Study Week 40)
Population: Safety Population: all participants (KRAS, BRAF, NRAS, and MEK1 mutation positive) that received at least one dose of study treatment, based on the actual treatment received if this differed from that to which the participant was randomized. Only participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP
Number analyzed (Participants) | 87 | 43
Participants
  Albumin, Increase to any G (IAG), n=86, 43 | 57 | 21
  Albumin, Increase to G3, n=86, 43 | 4 | 1
  Albumin, Increase to G4, n=86, 43 | 0 | 0
  ALKP, IAG, n=85, 43 | 26 | 3
  ALKP, Increase to G3, n =85, 43 | 2 | 1
  ALKP, Increase to G4, n=85, 43 | 0 | 0
  ALT, IAG, n=87, 43 | 32 | 7
  ALT, Increase to G3, n=87, 43 | 3 | 1
  ALT, Increase to G4, n=87, 43 | 0 | 0
  AST, IAG, n=86, 43 | 55 | 11
  AST, Increase to G3, n=86, 43 | 1 | 0
  AST, Increase to G4, n=86, 43 | 0 | 0
  Total bilirubin, IAG, n=85, 42 | 3 | 3
  Total bilirubin, Increase to G3, n=85, 42 | 0 | 0
  Total bilirubin, Increase to G4, n=85, 42 | 0 | 0
  Calcium (hypercalcemia), IAG, n =87, 43 | 9 | 3
  Calcium (hypercalcemia), Increase to G3, n=87, 43 | 0 | 0
  Calcium (hypercalcemia), Increase to G4, n=87, 43 | 0 | 0
  Calcium (hypocalcemia), IAG, n=87, 43 | 4 | 1
  Calcium (hypocalcemia), Increase to G3, n=87, 43 | 0 | 1
  Calcium (hypocalcemia), Increase to G4, n=87, 43 | 1 | 0
  Creatine kinase, IAG, n=1, 0 | 0 | 0
  Creatine kinase, Increase to G3, n=1, 0 | 0 | 0
  Creatine kinase, Increase to G4, n=1, 0 | 0 | 0
  Creatinine, IAG, n=87, 43 | 12 | 6
  Creatinine, Increase to G3, n=87, 43 | 3 | 1
  Creatinine, Increase to G4, n=87, 43 | 0 | 0
  Glucose (hyperglycemia), IAG, n=87, 43 | 47 | 24
  Glucose (hyperglycemia), Increase to G3, n=87, 43 | 5 | 2
  Glucose (hyperglycemia), Increase to G4, n=87, 43 | 0 | 0
  Glucose (hypoglycemia), IAG, n=87, 43 | 4 | 4
  Glucose (hypoglycemia), Increase to G3, n=87, 43 | 0 | 0
  Glucose (hypoglycemia), Increase to G4, n=87, 43 | 0 | 0
  Potassium (hyperkalemia), IAG, n=86, | 9 | 4
  Potassium (hyperkalemia), Increase to G3, n=86, 43 | 1 | 1
  Potassium (hyperkalemia), Increase to G4, n=86, 43 | 0 | 0
  Potassium (hypokalemia), IAG, n=86, 43 | 8 | 2
  Potassium (hypokalemia), Increase to G3, n=86, 43 | 0 | 0
  Potassium (hypokalemia), Increase to G4, n=86, 43 | 0 | 0
  Sodium (hypernatremia), IAG, n=87, 43 | 12 | 2
  Sodium (hypernatremia), Increase to G3, n=87, 43 | 0 | 0
  Sodium (hypernatremia), Increase to G4, n=87, 43 | 0 | 0
  Sodium (hyponatremia), IAG, n=87, 43 | 16 | 5
  Sodium (hyponatremia), Increase to G3, n=87, 43 | 2 | 1
  Sodium (hyponatremia), Increase to G4, n=87, 43 | 0 | 0

3. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline in the Indicated Clinical Chemistry Parameters: Crossover Phase
Description: Clinical chemistry parameters were summarized according to NCI CTCAE grade, version 4.0. Grade (G) 1, Mild; Grade 2, Moderate; Grade 3 (G3), Severe; Grade 4 (G4), Life-threatening or disabling; Grade 5, Death. Data are presented for only those parameters for which an increase to any grade, Grade 3, or Grade 4 occurred. Clinical chemistry parameters included: albumin, alkaline phosphatase (ALKP), alanine amino transferase (ALT), aspartate amino transferase (AST), total bilirubin, calcium (hypercalcemia), calcium (hypocalcemia), creatine kinase, creatinine, glucose (hyperglycemia), glucose (hypoglycemia), potassium (hyperkalemia), potassium (hypokalemia), sodium (hypernatremia), and sodium (hyponatremia). Worst-case on-therapy changes from Baseline were summarized. Worst-case on-therapy was defined using the on-therapy window and changes were indentified using both scheduled and unscheduled assessments.
Time Frame: Baseline; Days 1, 8, and 15 of Cycle 1; and Day 1 of every cycle thereafter until treatment discontinuation of the Crossover Phase (up to Study Week 19)
Population: Crossover Population: all participants who, at the point of disease progression during the Randomized Phase, elected to enter the crossover portion of the study. Only participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg in CP | Docetaxel 75 mg/m^2 in CP
Number analyzed (Participants) | 23 | 1
Participants
  Albumin, Increase to any G (IAG), n=23, 1 | 15 | 1
  Albumin, Increase to G3, n=23, 1 | 4 | 0
  Albumin, Increase to G4, n=23, 1 | 0 | 0
  ALKP, IAG, n=23, 1 | 10 | 0
  ALKP, Increase to G3, n =23, 1 | 1 | 0
  ALKP, Increase to G4, n=23, 1 | 0 | 0
  ALT, IAG, n=23, 1 | 7 | 0
  ALT, Increase to G3, n=23, 1 | 1 | 0
  ALT, Increase to G4, n=23, 1 | 0 | 0
  AST, IAG, n=23, 1 | 9 | 0
  AST, Increase to G3, n=23, 1 | 1 | 0
  AST, Increase to G4, n=23, 1 | 0 | 0
  Total bilirubin, IAG, n=22, 1 | 1 | 0
  Total bilirubin, Increase to G3, n=22, 1 | 0 | 0
  Total bilirubin, Increase to G4, n=22, 1 | 0 | 0
  Calcium (hypercalcemia), IAG, n =23, 1 | 1 | 0
  Calcium (hypercalcemia), Increase to G3, n=23, 1 | 0 | 0
  Calcium (hypercalcemia), Increase to G4, n=23, 1 | 0 | 0
  Calcium (hypocalcemia), IAG, n=23, 1 | 0 | 0
  Calcium (hypocalcemia), Increase to G3, n=23, 1 | 0 | 0
  Calcium (hypocalcemia), Increase to G4, n=23, 1 | 0 | 0
  Creatine kinase, IAG, n=1, 0 | 1 | 0
  Creatine kinase, Increase to G3, n=1, 0 | 0 | 0
  Creatine kinase, Increase to G4, n=1, 0 | 0 | 0
  Creatinine, IAG, n=23, 1 | 3 | 0
  Creatinine, Increase to G3, n=23, 1 | 0 | 0
  Creatinine, Increase to G4, n=23, 1 | 0 | 0
  Glucose (hyperglycemia), IAG, n=23, 1 | 10 | 0
  Glucose (hyperglycemia), Increase to G3, n=23, 1 | 0 | 0
  Glucose (hyperglycemia), Increase to G4, n=23, 1 | 0 | 0
  Glucose (hypoglycemia), IAG, n=23, 1 | 1 | 0
  Glucose (hypoglycemia), Increase to G3, n=23, 1 | 0 | 0
  Glucose (hypoglycemia), Increase to G4, n=23, 1 | 0 | 0
  Potassium (hyperkalemia), IAG, n=23, 1 | 3 | 0
  Potassium (hyperkalemia), Increase to G3, n=23, 1 | 1 | 0
  Potassium (hyperkalemia), Increase to G4, n=23, 1 | 0 | 0
  Potassium (hypokalemia), IAG, n=23, 1 | 1 | 0
  Potassium (hypokalemia), Increase to G3, n=23, 1 | 0 | 0
  Potassium (hypokalemia), Increase to G4, n=23, 1 | 0 | 0
  Sodium (hypernatremia), IAG, n=23, 1 | 1 | 0
  Sodium (hypernatremia), Increase to G3, n=23, 1 | 0 | 0
  Sodium (hypernatremia), Increase to G4, n=23, 1 | 0 | 0
  Sodium (hyponatremia), IAG, n=23, 1 | 3 | 0
  Sodium (hyponatremia), Increase to G3, n=23, 1 | 2 | 0
  Sodium (hyponatremia), Increase to G4, n=23, 1 | 0 | 0

4. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline in the Indicated Hematology Parameters: Randomized Phase
Description: Hematology parameters were summarized according to NCI CTCAE grade, version 4.0. Grade (G) 1, Mild; Grade 2, Moderate; Grade 3 (G3), Severe; Grade 4 (G4), Life-threatening or disabling; Grade 5, Death. Data are presented for only those parameters for which an increase to any G (IAG), G3, or G4 occurred. Hematology parameters included: haemoglobin (increased [inc]), haemoglobin (anemia), lymphocyte count (ct) (inc), lymphocyte ct (decreased [dec]), total absolute neutrophil count (ANC), platelet ct, and white blood cell count (WBC). Worst-case on-therapy changes from Baseline were summarized. Worst-case on-therapy was defined using the on-therapy window and changes were indentified using both scheduled and unscheduled assessments.
Time Frame: as for outcome 2
Population: Safety Population. Only participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP
Number analyzed (Participants) | 87 | 43
Participants
  Haemoglobin (inc), IAG, n=87, 43 | 0 | 0
  Haemoglobin (inc), Increase to G3, n=87, 43 | 0 | 0
  Haemoglobin (inc), Increase to G4, n=87, 43 | 0 | 0
  Haemoglobin (anemia), IAG, n=86, 43 | 34 | 27
  Haemoglobin (anemia), Increase to G3, n=86, 43 | 8 | 3
  Haemoglobin (anemia), Increase to G4, n=86, 43 | 0 | 0
  Lymphocyte ct (inc), IAG, n=86, 43 | 9 | 2
  Lymphocyte ct (inc), Increase to G3, n=86, 43 | 1 | 0
  Lymphocyte ct (inc), Increase to G4, n=86, 43 | 0 | 0
  Lymphocyte ct (dec), IAG, n=85, 43 | 18 | 19
  Lymphocyte ct (dec), Increase to G3, n=85, 43 | 4 | 2
  Lymphocyte ct (dec), Increase to G4, n=85, 43 | 0 | 0
  ANC, IAG, n=86, 43 | 5 | 34
  ANC, Increase to G3, n=86, 43 | 0 | 13
  ANC, Increase to G4, n=86, 43 | 0 | 13
  Platelet ct, IAG, n=87, 43 | 15 | 3
  Platelet ct, Increase to G3, n=87, 43 | 0 | 0
  Platelet ct, Increase to G4, n=87, 43 | 0 | 0
  WBC, IAG, n=87, 43 | 5 | 33
  WBC, Increase to G3, n=87, 43 | 0 | 17
  WBC, Increase to G4, n=87, 43 | 1 | 0

5. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline in the Indicated Hematology Parameters: Crossover Phase
Description: as for outcome 4
Time Frame: as for outcome 3
Population: Crossover Population. Only participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg in CP | Docetaxel 75 mg/m^2 in CP
Number analyzed (Participants) | 23 | 1
Participants
  Haemoglobin (inc), IAG, n=23, 1 | 0 | 0
  Haemoglobin (inc), Increase to G3, n=23, 1 | 0 | 0
  Haemoglobin (inc), Increase to G4, n=23, 1 | 0 | 0
  Haemoglobin (anemia), IAG, n=23, 1 | 12 | 0
  Haemoglobin (anemia), Increase to G3, n=23, 1 | 2 | 0
  Haemoglobin (anemia), Increase to G4, n=23, 1 | 0 | 0
  Lymphocyte ct (inc), IAG, n=23, 1 | 1 | 0
  Lymphocyte ct (inc), Increase to G3, n=23, 1 | 0 | 0
  Lymphocyte ct (inc), Increase to G4, n=23, 1 | 0 | 0
  Lymphocyte ct (dec), IAG, n=23, 1 | 3 | 0
  Lymphocyte ct (dec), Increase to G3, n=23, 1 | 0 | 0
  Lymphocyte ct (dec), Increase to G4, n=23, 1 | 0 | 0
  ANC, IAG, n=19, 0 | 0 | 0
  ANC, Increase to G3, n=19, 0 | 0 | 0
  ANC, Increase to G4, n=19, 0 | 0 | 0
  Platelet ct, IAG, n=23, 1 | 4 | 0
  Platelet ct, Increase to G3, n=23, 1 | 0 | 0
  Platelet ct, Increase to G4, n=23, 1 | 0 | 0
  WBC, IAG, n=23, 1 | 0 | 0
  WBC, Increase to G3, n=23, 1 | 0 | 0
  WBC, Increase to G4, n=23, 1 | 0 | 0

6. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline With Respect to Normal Ranges in the Indicated Clinical Chemistry Parameters: Randomized Phase
Description: Data are presented for only those clinical chemistry parameters for which the following worst-case on-therapy changes from Baseline with respect to the normal range were observed: decrease to low, change to normal (CTN) or no change, or increase to high. Clinical chemistry parameters included: lactate dehydrogenase, total protein, and urea/blood urea nitrogen (BUN). Worst-case on-therapy changes from Baseline were summarized. Worst-case on-therapy was defined using the on-therapy window and changes were indentified using both scheduled and unscheduled assessments. Normal ranges for each parameter may vary depending on the laboratory (central versus local) and the participant (age, gender, etc.).
Time Frame: as for outcome 2
Population: Safety Population. Only participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP
Number analyzed (Participants) | 87 | 43
Participants
  Lactate dehydrogenase, Decrease to low, n=87, 43 | 1 | 0
  Lactate dehydrogenase, CTN or no change, n=87, 43 | 40 | 23
  Lactate dehydrogenase, Increase to high, n=87, 43 | 46 | 20
  Total Protein, Decrease to low, n=86, 43 | 31 | 12
  Total Protein, CTN or no change, n=86, 43 | 55 | 31
  Total Protein, Increase to high, n=86, 43 | 1 | 0
  Urea/BUN, Decrease to low, n=87, 43 | 0 | 0
  Urea/BUN, CTN or no change, n=87, 43 | 62 | 34
  Urea/BUN, Increase to high, n=87,43 | 25 | 9

7. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline With Respect to Normal Ranges in the Indicated Clinical Chemistry Parameters: Crossover Phase
Description: as for outcome 6
Time Frame: as for outcome 3
Population: Crossover Population. Only participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg in CP | Docetaxel 75 mg/m^2 in CP
Number analyzed (Participants) | 23 | 1
Participants
  Lactate dehydrogenase, Decrease to low | 0 | 0
  Lactate dehydrogenase, CTN or no change | 15 | 1
  Lactate dehydrogenase, Increase to high | 8 | 0
  Total Protein, Decrease to low | 15 | 0
  Total Protein, CTN or no change | 8 | 1
  Total Protein, Increase to high | 0 | 0
  Urea/BUN, Decrease to low | 0 | 0
  Urea/BUN, CTN or no change | 18 | 1
  Urea/BUN, Increase to high | 5 | 0

8. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline With Respect to Normal Ranges in the Indicated Hematology Parameters: Randomized Phase
Description: Data are presented for only those hematology parameters for which the following worst-case on-therapy changes from Baseline with respect to the normal range were observed: decrease to low, change to normal (CTN) or no change, or increase to high. Hematology parameters included: atypical lymphs, atypical lymphs (percentage [%]), basophils, eosinophils, metamyelocytes, monocytes, myelocytes, neutrophil bands (%). Worst-case on-therapy changes from Baseline were summarized. Worst-case on-therapy was defined using the on-therapy window and changes were indentified using both scheduled and unscheduled assessments. Normal ranges for each parameter may vary depending on the laboratory (central versus local) and the participant (age, gender, etc.).
Time Frame: as for outcome 2
Population: Safety Population. Only participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP
Number analyzed (Participants) | 86 | 43
Participants
  Atypical lymphs, Decrease to low, n=0, 3 | 0 | 0
  Atypical lymphs, CTN or no change, n=0, 3 | 0 | 0
  Atypical lymphs, Increase to high, n=0, 3 | 0 | 3
  Atypical lymphs (%), Decrease to low, n =0, 3 | 0 | 0
  Atypical lymphs (%), CTN or no change, n=0, 3 | 0 | 0
  Atypical lymphs (%), Increase to high, n=0, 3 | 0 | 3
  Basophils, Decrease to low, n=86, 43 | 0 | 0
  Basophils, CTN or no change, n=86, 43 | 82 | 41
  Basophils, Increase to high, n=86,43 | 4 | 2
  Eosinophils, Decrease to low, n=86, 43 | 1 | 1
  Eosinophils, CTN or no change, n=86, 43 | 77 | 42
  Eosinophils, Increase to high, n=86, 43 | 9 | 0
  Metamyelocytes, Decrease to low, n=1, 7 | 0 | 0
  Metamyelocytes, CTN or no change, n=1, 7 | 0 | 0
  Metamyelocytes, Increase to high, n=1, 7 | 1 | 7
  Monocytes, Decrease to low, n=86, 43 | 3 | 20
  Monocytes, CTN or no change, n=86, 43 | 78 | 18
  Monocytes, Increase to high, n=86, 43 | 5 | 9
  Myelocytes, Decrease to low, n=1, 9 | 0 | 0
  Myelocytes, CTN or no change, n=1, 9 | 0 | 1
  Myelocytes, Increase to high, n=1, 9 | 1 | 8
  Neutrophil Bands (%), Decrease to low, n=1, 4 | 0 | 0
  Neutrophil Bands (%), CTN or no change, n=1, 4 | 1 | 3
  Neutrophil Bands (%), Increase to high, n=1, 4 | 0 | 1

9. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline With Respect to Normal Ranges in the Indicated Hematology Parameters: Crossover Phase
Description: Data are presented for only those hematology parameters for which the following worst-case on-therapy changes from Baseline with respect to the normal range were observed: decrease to low, change to normal (CTN) or no change, or increase to high. Hematology parameters included: atypical lymphs, atypical lymphs (percentage [%]), basophils, eosinophils, metamyelocytes, monocytes, and myelocytes. Worst-case on-therapy changes from Baseline were summarized. Worst-case on-therapy was defined using the on-therapy window and changes were indentified using both scheduled and unscheduled assessments. Normal ranges for each parameter may vary depending on the laboratory (central versus local) and the participant (age, gender, etc.).
Time Frame: as for outcome 3
Population: Crossover Population. Only participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg in CP | Docetaxel 75 mg/m^2 in CP
Number analyzed (Participants) | 23 | 1
Participants
  Atypical lymphs, Decrease to low, n=3, 1 | 0 | 0
  Atypical lymphs, CTN or no change, n=3, 1 | 1 | 0
  Atypical lymphs, Increase to high, n=3, 1 | 2 | 1
  Atypical lymphs (%), Decrease to low, n=3, 1 | 0 | 0
  Atypical lymphs (%), CTN or no change, n=3, 1 | 1 | 0
  Atypical lymphs (%), Increase to high, n=3, 1 | 2 | 1
  Basophils, Decrease to low, n=23, 1 | 0 | 0
  Basophils, CTN or no change, n=23, 1 | 23 | 1
  Basophils, Increase to high, n=23, 1 | 0 | 0
  Eosinophils, Decrease to low, n=23, 1 | 0 | 0
  Eosinophils, CTN or no change, n=23, 1 | 23 | 1
  Eosinophils, Increase to high, n=23, 1 | 0 | 0
  Metamyelocytes, Decrease to low, n=1, 1 | 0 | 0
  Metamyelocytes, CTN or no change, n=1, 1 | 0 | 0
  Metamyelocytes, Increase to high, n=1, 1 | 1 | 1
  Monocytes, Decrease to low, n=23, 1 | 1 | 0
  Monocytes, CTN or no change, n=23, 1 | 20 | 0
  Monocytes, Increase to high, n=23, 1 | 2 | 1
  Myelocytes, Decrease to low, n=3, 1 | 0 | 0
  Myelocytes, CTN or no change, n=3, 1 | 0 | 0
  Myelocytes, Increase to high, n=3, 1 | 3 | 1

10. Secondary Outcome: Number of Participants With Any Serious Adverse Event (SAE) or Non-serious Adverse Event (AE): Randomized Phase
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. Medical or scientific judgment should have been exercised in deciding whether reporting was appropriate in other situations. Refer to the general Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From randomization until 30 days following discontinuation of study treatment regardless of initiation of a new cancer therapy or transfer to hospice (maximum of 19 months)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP
Number analyzed (Participants) | 87 | 43
Participants
  Any AE | 87 | 43
  Any SAE | 32 | 9

11. Secondary Outcome: Number of Participants With Any SAE or Non-serious AE: Crossover Phase
Description: as for outcome 10
Time Frame: From the date of the first dose of study treatment in the Crossover Phase until 30 days following discontinuation of study treatment regardless of initiation of a new cancer therapy or transfer to hospice (maximum of 12 months)
Population: Crossover Population
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg in CP | Docetaxel 75 mg/m^2 in CP
Number analyzed (Participants) | 23 | 2
Participants
  Any AE | 22 | 2
  Any SAE | 12 | 1

12. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP): Randomized Phase
Description: Systolic and diastolic blood pressure were measured at the following scheduled time points: Baseline; Days 1, 8, and 15 of Cycle 1 (Study Week 1); and Day 1 of every cycle thereafter until treatment discontinuation. The worst-case on-therapy was determined using both scheduled and unscheduled assessments during the on-therapy period. Change from Baseline was calculated as the value at post-Baseline time point minus the value at Baseline.
Time Frame: as for outcome 2
Population: Safety Population. Only participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP
Number analyzed (Participants) | 87 | 43
millimeters of mercury (mmHg)
  SBP, Worst-case on-therapy | 13.5 (16.63) | 3.1 (13.71)
  DBP, Worst-case on-therapy | 10.7 (9.95) | 2.5 (7.34)

13. Secondary Outcome: Change From Baseline in SBP and DBP: Crossover Phase
Description: Systolic and diastolic blood pressure were measured at the following scheduled time points: Baseline; Days 1, 8, and 15 of Cycle 1 (Study Week 1); and Day 1 of every cycle therafter until treatment discontinuation. The worst-case on-therapy was determined using both scheduled and unscheduled assessments during the on-therapy period. Change from Baseline was calculated as the value at post-Baseline time point minus the value at Baseline.
Time Frame: as for outcome 3
Population: Crossover Population. Only participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | GSK1120212 2 mg in CP | Docetaxel 75 mg/m^2 in CP
Number analyzed (Participants) | 23 | 1
mmHg
  SBP, Worst-case on-therapy | 8.7 (15.95) | -15.0 (NA) — Only one participant was analyzed in this treatment arm at this time point; therefore the standard deviation cannot be calculated.
  DBP, Worst-case on-therapy | 8.3 (12.28) | -12.0 (NA) — Only one participant was analyzed in this treatment arm at this time point; therefore the standard deviation cannot be calculated.

14. Secondary Outcome: Change From Baseline in Heart Rate: Randomized Phase
Description: Heart rate was measured at the following scheduled time points: Baseline; Days 1, 8, and 15 of Cycle 1 (Study Week 1); and Day 1 of every cycle therafter until treatment discontinuation.The worst-case on-therapy was determined using both scheduled and unscheduled assessments during the on-therapy period. Change from Baseline was calculated as the value at post-Baseline time point minus the value at Baseline.
Time Frame: as for outcome 2
Population: Safety Population. Only participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP
Number analyzed (Participants) | 87 | 43
Beats per minute | 10.4 (14.23) | 13.2 (9.31)

15. Secondary Outcome: Change From Baseline in Heart Rate: Crossover Phase
Description: as for outcome 14
Time Frame: as for outcome 3
Population: Crossover Population. Only participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK1120212 2 mg in CP | Docetaxel 75 mg/m^2 in CP
Number analyzed (Participants) | 23 | 1
Beats per minute | 8.5 (11.46) | 5.0 (NA) — Only one participant was analyzed in this treatment arm at this time point; therefore the standard deviation cannot be calculated.

16. Secondary Outcome: Number of Participants With a Best Response of Either a Complete Response (CR) or Partial Response (PR) as Assessed by the Investigator: Randomized Phase
Description: Response was assessed by the investigator according to RECIST, version 1.1, using confirmed and unconfirmed responses. Responders were defined as participants achieving either a CR (disappearance of all target and non-target lesions; any pathological lymph nodes must be <10 millimeters [mm] in the short axis; without the appearance of new lesions) or PR (at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]). Participants with unknown or missing response were treated as non-responders.
Time Frame: From randomization until the first documented evidence of a CR or PR (maximum of 10.2 months)
Population: MITT Population
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP
Number analyzed (Participants) | 86 | 43
Participants
  CR | 0 | 0
  PR | 10 | 5

17. Secondary Outcome: Number of Participants With a Best Response of Either a CR or PR as Assessed by the Investigator: Crossover Phase
Description: as for outcome 16
Time Frame: From the date of the first dose of study treatment in the Crossover Phase until the first documented evidence of a CR or PR (maximum of 4 months)
Population: Crossover Population
Measure: Number; unit: Participants
Arm/Group | GSK1120212 2 mg in CP | Docetaxel 75 mg/m^2 in CP
Number analyzed (Participants) | 23 | 2
Participants
  CR | 0 | 0
  PR | 1 | 0

18. Secondary Outcome: Duration of Response (DOR) as Assessed by the Investigator: Randomized Phase
Description: DOR was assessed by the investigator for participants with CR (disappearance of all target and non-target lesions; any pathological lymph nodes must be <10 mm in the short axis; without the appearance of new lesions) or PR (at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]). DOR is defined as the time from the first documented evidence of CR or PR until the earliest date of documented radiological progression or death due to any cause. PD is defined as at least a 20% increase in the sum of the diameters (SD) of target lesions with an absolute increase of at least 5 millimeters (mm) or the appearance of at least 1 new lesion, or the worsening of non-target lesions significant enough to require study treatment discontinuation.
Time Frame: Time from the first documented evidence of CR or PR until the earliest date of documented radiological progression or death due to any cause (maximum of 10.2 months)
Population: MITT Population. Only participants who achieved a CR or PR were analyzed for duration of response.
Measure: Mean (95% Confidence Interval); unit: Weeks
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP
Number analyzed (Participants) | 10 | 5
Weeks | 6.7 [2.7 to NA] — There were a limited number of participants with a CR or PR who later progressed or died; therefore, the upper limit (UL) of the CI could not be estimated. | 12.4 [7.1 to 17.3]

19. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the interval of time between the date of randomization and the date of death due to any cause. For participants who did not die, OS was censored at the date of last contact.
Time Frame: Time interval between the date of randomization and the date of death due to any cause (maximum of 22 months)
Population: MITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP
Number analyzed (Participants) | 86 | 43
Months | 8.1 [6.8 to 10.0] | 9.9 [5.0 to NA] — Statistics for the median is missing because an insufficient number of participants reached the milestone, making calculation of this statistic inappropriate or impossible.

20. Secondary Outcome: GSK1120212 Plasma Pharmacokinetic (PK) Concentration
Description: Blood samples for PK analysis of GSK1120212 were collected at the following time points: Cycle 1 (Study Day 15), Cycle 2 (Study Day 22), Cycle 3 (Study Day 43), and Cycle 4 (Study Day 64). Post-dose PK samples collected on Day 15 of Cycle 1 occurred at least 1 hour apart. Participants were instructed to withhold the dose of GSK1120212 until after blood for PK samples had been drawn. Pre-dose samples were taken 15 minutes or less prior to taking the next dose (i.e., trough).
Time Frame: Day 15 of Cycle 1: pre-dose; 0.5-2 hours, 2-4 hours, and 4-8 hours post-dose; Day 1 of Cycle 2, Cycle 3 and Cycle 4: pre-dose
Population: PK Population. Only participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms (ng)/milliliter (mL)
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP
Number analyzed (Participants) | 80 | 0
Nanograms (ng)/milliliter (mL)
  Cycle 1, Day 15, pre-dose, n=80 | 16.1 (5.31) |
  Cycle 1, Day 15, 0.5-2 hours post-dose, n=78 | 21.5 (8.59) |
  Cycle 1, Day 15, 2-4 hours post-dose, n=77 | 29.7 (22.9) |
  Cycle 1, Day 15, 4-8 hours post-dose, n=78 | 24.8 (7.80) |
  Cycle 2, Day 1, pre-dose, n=75 | 16.7 (6.95) |
  Cycle 3, Day 1, pre-dose, n=60 | 12.9 (7.19) |
  Cycle 4, Day 1, pre-dose, n=38 | 13.9 (6.49) |

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) and non-serious AEs were collected from the first dose of study treatment until 30 days following discontinuation of study treatment regardless of initiation of a new cancer therapy (maximum of 19 months).
Description: SAEs and non-serious AEs were collected in members of the Safety Population (all participants who received at least one dose of study treatment) and the Crossover Population (participants who, at the point of disease progression during the Randomized Phase, elected to enter the crossover portion of the study).
Groups:
- GSK1120212 2 mg in RP: Participants received GSK1120212 2 milligrams (mg) orally once daily continuously in the Randomized Phase (RP). Participants continued treatment until disease progression, death, or unacceptable adverse events were experienced.
- Docetaxel 75 mg/m^2 in RP: Participants received docetaxel 75 mg per meters squared (m^2) intravenously (IV) every 3 weeks in the RP. Participants continued treatment on a 21-day cycle until disease progression, death, or unacceptable adverse events were experienced.
- GSK1120212 2 mg in CP: Participants who experienced disease progression in the RP were given the option of crossing over to GSK1120212 2 mg and continuing in the Cross-over Phase (CP).
- Docetaxel 75 mg/m^2 in CP: Participants who experienced disease progression in the RP were given the option of crossing over to docetaxel 75 mg/m^2 and continuing in the CP.
Arm/Group | GSK1120212 2 mg in RP | Docetaxel 75 mg/m^2 in RP | GSK1120212 2 mg in CP | Docetaxel 75 mg/m^2 in CP
Serious Adverse Events (participants affected / at risk) | 32/87 | 9/43 | 12/23 | 1/2
Other Adverse Events (participants affected / at risk) | 87/87 | 43/43 | 20/23 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1120212 2 mg in RP (N=87) | Docetaxel 75 mg/m^2 in RP (N=43) | GSK1120212 2 mg in CP (N=23) | Docetaxel 75 mg/m^2 in CP (N=2)
Pneumonia (Infections and infestations) | 6 | 1 | 2 | 0
Sepsis (Infections and infestations) | 4 | 1 | 2 | 0
Pneumocystis jiroveci infection (Infections and infestations) | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Sigmoiditis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 3 | 1 | 0 | 0
Oedema (General disorders) | 2 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 2 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 2 | 0 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1120212 2 mg in RP (N=87) | Docetaxel 75 mg/m^2 in RP (N=43) | GSK1120212 2 mg in CP (N=23) | Docetaxel 75 mg/m^2 in CP (N=2)
Rash (Skin and subcutaneous tissue disorders) | 50 | 6 | 7 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 17 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 2 | 3 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 11 | 2 | 2 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 8 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0
Fatigue (General disorders) | 24 | 12 | 0 | 0
Asthenia (General disorders) | 20 | 11 | 4 | 1
Oedema peripheral (General disorders) | 19 | 5 | 7 | 0
Pyrexia (General disorders) | 15 | 4 | 3 | 0
Mucosal inflammation (General disorders) | 6 | 6 | 0 | 0
Face oedema (General disorders) | 6 | 2 | 0 | 0
Oedema (General disorders) | 6 | 1 | 0 | 0
Chills (General disorders) | 6 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 44 | 9 | 11 | 1
Nausea (Gastrointestinal disorders) | 30 | 12 | 5 | 0
Constipation (Gastrointestinal disorders) | 18 | 7 | 5 | 0
Vomiting (Gastrointestinal disorders) | 20 | 5 | 5 | 0
Dry mouth (Gastrointestinal disorders) | 13 | 1 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 9 | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 8 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 3 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 7 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 7 | 6 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 30 | 8 | 2 | 0
Hypotension (Vascular disorders) | 9 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 21 | 7 | 5 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 | 1 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 18 | 8 | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 15 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 5 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 10 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 6 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 7 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 7 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 3 | 0 | 0
Ejection fraction decreased (Investigations) | 5 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 3 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 5 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 9 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 5 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 9 | 0 | 0
Confusional state (Psychiatric disorders) | 5 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 3 | 1 | 1
Paronychia (Infections and infestations) | 7 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 3 | 3 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Headache (Nervous system disorders) | 5 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.